CLINICAL TRIAL: NCT06322862
Title: Intraoperative Intestinal Perfusion Assessment by Fluorescence Angiography in Emergency Surgery
Brief Title: FLuorescence Guided Assessment of Mesenteric Ischemia in Emergency Surgery
Acronym: FLAMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Patrick Achiam, Professor, MD, PhD, DMSc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-23042430
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Bowel; Ischemic, Acute
Keywords: indocyanine green; perfusion assessment; acute care surgery
MeSH Terms: conditions — Ischemia | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Other)
  Interventions: Other: Indocyanine green

INTERVENTIONS:
Other: Indocyanine green — Intraoperative perfusion assessment with ICG Fluorescence Angiography (ICG-FA) in standard approved doses

SUMMARY:
This is a prospective, multicentre, non-randomized cohort study using real-time intraoperative visualization of bowel perfusion by indocyanine green (ICG) in all-cause bowel ischemia.

At intraoperative finding of bowel ischemia, the initial intraoperative plan is noted and resection margins marked with a steril pen. A fluorescence angiography will be performed and the surgeon will note whether the suspected ischemic bowel is perfused, whether there is a change in the resection margins in centimeters, and if the intraoperative plan has changed. If resection is indicated and the strategy of choice is an anastomosis, a renewed fluorescence angiography will be performed to assess anastomotic perfusion.

DETAILED DESCRIPTION:
Fluorescence guided-surgery utilises the fluorescent property of a fluorophore, indocyanine green (ICG), injected intravenously to assess perfusion and viability of the bowel.

This study aims to evaluate the usability and feasibility of ICG to assess bowel viability in an emergency abdominal surgery setting where all-cause bowel ischemia is suspected and intraoperatively present. The investigators aim to evaluate whether ICG fluorescence angiography contributes as an intraoperative aid and changes the intraoperative strategy.

The investigators hypothesize that ICG is a safe and reliable aid in intraoperative decision-making regarding mesenteric ischemia. It may lead to an increasing number of one-step definitive procedures with vital resection margins, primary anastomosis and reducing stomas, and second-look procedures.

In this prospective, non-randomized cohort study bowel viability will be assessed using intraoperative real-time visualization by performing an ICG-fluorescence angiography when there is intraoperative finding of bowel ischemia.

Intraoperatively, ICG (Verdye, Diagnostic Green GmbH 25 mg vials) are dissolved with 5 ml sterile water obtaining a concentration of 5 mg/ml. 0,2mg/kg will be administered intravenously at one to two steps of perfusion assessment.

Initially, the surgeon notes the intended intraoperative plan before fluorescing and if resection is deemed necessary, the resection margins will be marked with a sterile pen.

The perfusion assessment with ICG is then performed and perfusion of the suspected ischemic bowel is noted, along with any change in intended resection margins and intraoperative plan. If an anastomosis is performed, a renewed perfusion assessment is performed. The perfusion assessment will be recorded.

Postoperatively, a subgroup of suitable perfusion assessment recordings will be subject to quantification software using software developed and validated by the investigators (q-ICG).

The trial follows regulations for research in emergency settings and a written and oral informed consent will be obtained from the participant or the participants next of kin and a trial guardian, postoperatively.

Intra- and postoperative clinical data will be collected, including choice of strategy, anastomotic leaks, 30- and 90- day complications, and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years of age
* Acute physiologic derangement and suspected of having bowel ischemia
* Intraoperative finding of all-cause bowel ischemia with subsequent acute physiologic derangement

Exclusion Criteria:

* Allergy toward; iodine, indocyanine green, or shellfish
* Liver insufficiency
* Thyrotoxicosis
* Pregnancy or lactation
* Permanently legally incompetent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change of strategy | Assessed at day 30 and 90 after surgery
  Change of intraoperative strategy due to ICG fluorescence angiography. Intraoperatively, a nurse will record the initial strategy, indication of resection in centimeters, before and after ICG angiography, and note whether there has been a change in strategy, and how.

SECONDARY OUTCOMES:
Anastomosis | Assessed at day 30 and 90 after surgery
  Number of anastomoses established in ICG-perfused bowel segments
Quantification using q-ICG | 30 months
  A posthoc perfusion quantification using q-ICG software
Stomas | Assessed at day 30 and 90 after surgery
  Number of cases where stoma was the preferred strategy
Second-look | Assessed at day 30 and 90 after surgery
  Number of cases where second-look following bowel discontinuation, was the preferred strategy
Anastomotic leaks | Assessed at day 30 and 90 after surgery
  Cases of anastomotic leaks postoperatively
Postoperative medical complications | Assessed at day 30 and 90 after surgery
  Stratified by type and severity (Comprehensive Complication Index)
Postoperative surgical complications | Assessed at day 30 and 90 after surgery
  Stratified by type and severity (Comprehensive Complication Index)
Mortality | 90 days
  30- and 90-day mortality rates

CONTACTS AND LOCATIONS:
Overall Officials: Sermed Ellebæk Nicolae, MD, PhDstudent, Principal Investigator — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Department of Organ Surgery and Transplantation, Copenhagen, Capital Region
  - Department of Surgery, Bispebjerg Hospital, Bispebjerg
  - Department of Surgery, Herlev Hospital, Herlev
  - Department of Surgery, Nordsjællands Hospital, Hillerød
  - Department of Surgery, Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No